CLINICAL TRIAL: NCT00428090
Title: A 24-week, Double-blind, Double-dummy, Randomized, Parallel-group Study to Investigate the Effects of Rosiglitazone (Extended Release Tablets), Donepezil, and Placebo as Monotherapy on Cognition and Overall Clinical Response in APOE ε4-stratified Subjects With Mild to Moderate Alzheimer's Disease. (REFLECT-1)
Brief Title: Rosiglitazone (Extended Release Tablets) As Monotherapy In Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105640
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer's Disease
Keywords: apolipoprotein E; monotherapy; cognition; mild; rosiglitazone; Alzheimer's disease; moderate
MeSH Terms: conditions — Alzheimer Disease; Lymphoma, Follicular | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone (Experimental): XR (extended release) oral tablets
  Interventions: Drug: Rosiglitazone
- Placebo (Other): Placebo (Double-Dummy to Match)
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — XR (extended release) oral tablets

SUMMARY:
Rosiglitazone (RSG) has been tested and is approved as a treatment for type II diabetes mellitus, a disease that occurs when the body ineffectively uses glucose. RSG XR, the investigational drug, is an extended-release form of RSG. This study tests whether RSG XR safely provides benefit to people with mild to moderate Alzheimer's disease (AD). RSG XR is a new approach to AD therapy and this study tests whether one's genes alter the effectiveness of RSG XR. Glucose is used by cells to make energy that they need to live. Changes in the ability of cells to use of glucose can lead to diseases like diabetes. Glucose levels may be lower in the brains of AD patients, and their brain cells may also use glucose less well than in unaffected people. The proper function of brain cells may be critical to memory and thought. If brain cells use glucose poorly, this might impact AD. Drugs that help brain cells properly use glucose may help a person maintain normal memory and thinking. Data suggesting that RSG may help AD patients was first seen in a small study at the Univ. of Washington and then from a larger international GSK study. In the first study, those receiving RSG once daily for 6 months scored better on 3 tests of memory and thought than those who did not receive RSG. In the GSK study, those that benefited most from therapy with RSG XR had a specific genetic pattern. They lacked the gene that caused them to produce apolipoprotein E e4 (APOE e4). Subjects who have the APOE e4 gene may have two copies, one from each parent, or they may have only one APOE e4 gene meaning that they inherited either the APOE e2 or APOE e3 version of the gene from one parent. Subjects with one copy of the APOE e4 gene remained fairly stable while those with two copies of APOE e4 continued to worsen during the 6-month treatment. This study will directly test the effect of RSG XR on people who either have or lack the APOE e4 gene.

DETAILED DESCRIPTION:
A 24-week, double-blind, double-dummy, randomized, parallel-group study to investigate the effects of rosiglitazone (extended release tablets), donepezil, and placebo as monotherapy on cognition and overall clinical response in APOE e4-stratified subjects with mild to moderate Alzheimer's disease. (REFLECT-1)

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of probable Alzheimer's Disease (AD).
* MMSE score 10 to 23
* Has not taken an approved AD therapy in last 30 days.
* No previous hypersensitivity/intolerance to AChEIs
* Have a regular caregiver.

Exclusion criteria:

* Diagnosis of vascular dementia.
* Type I or secondary diabetes mellitus.
* Type II diabetes mellitus treated with insulin, sulfonylurea or glipizide.
* History or evidence of congestive heart failure, clinically significant peripheral edema or anemia.
* History of significant psychiatric illness, major depressive disorder or current depression needing initiation of treatment.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2007-02-27; Primary Completion 2008-09-01 (Actual); Study Completion 2008-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (109):
- United States (37):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Reseda, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Destin, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Sunrise, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Kenilworth, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Jenkintown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, DeSoto, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Middleton, Wisconsin
- Austria (4):
  - GSK Investigational Site, Graz-Eggenberg
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Vienna
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Chile (4):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- China (4):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- Croatia (2):
  - GSK Investigational Site, Dubrovnik
  - GSK Investigational Site, Zagreb
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (25):
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Günzburg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Baesweiler, North Rhine-Westphalia
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Jülich, North Rhine-Westphalia
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Itzehoe, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Gera, Thuringia
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Melíssia
  - GSK Investigational Site, Thessaloniki
- Hungary (5):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szeged
- India (3):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Tirupati
- Mexico (3):
  - GSK Investigational Site, Saltillo, Coahuila
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- GSK Investigational Site, Auckland, New Zealand
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- GSK Investigational Site, Lima, Peru
- Philippines (2):
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon City
- Puerto Rico (2):
  - GSK Investigational Site, Cabo Rojo, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Korea (2):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
- United Kingdom (3):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Derriford, Plymouth
  - GSK Investigational Site, West of Scotland Science Park, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gold M, Alderton C, Zvartau-Hind M, Egginton S, Saunders AM, Irizarry M, Craft S, Landreth G, Linnamagi U, Sawchak S. Rosiglitazone monotherapy in mild-to-moderate Alzheimer's disease: results from a randomized, double-blind, placebo-controlled phase III study. Dement Geriatr Cogn Disord. 2010;30(2):131-46. doi: 10.1159/000318845. Epub 2010 Aug 21. PMID 20733306
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 105640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105640 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) were enrolled across 134 centres Austria, Bulgaria, Chile, China, Crotia, Estonia, Germany, Greece, Hungry, Korea, Mexico, New Zealand, Pakistan, Peru, Philippines, Puerto Rico, Russia, the United Kingdom and the United States from February 2007 to September 2008. The total study duration was 30 weeks (W).
Pre-assignment Details: Total of 639 par. were screened out of which 581 were randomized and 58 were placebo run-in failures. Analysis population included 579 par. of 581 randomized participants as 2 par. did not take study drug: 1 from placebo and 1 from donepezil arm.
Groups:
- Placebo: Par. in this arm received RSG placebo tablet along with dummy donepezil capsule once daily for 24W. For par. in this arm, the dosage were remain constant throughout the 24W treatment period. Study treatment were taken in the evening with or without food.
- RSG XR 2 mg: Par. in this arm received rosiglitazone extended release (RSGXR) 2 milligram (mg) tablet along with dummy donepezil capsule once daily for 24W. For par. in this arm, the dosage were remain constant throughout the 24W treatment period. Study treatment were taken in the evening with or without food.
- RSG XR 8 mg: Par. in this arm received RSGXR 4 mg tablet along with dummy donepezil capsule once daily for the first 4W of treatment. From Visit 4 (W4) onwards, these par. received 8 mg RSGXR tablet along with dummy donepezil capsule once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
- Donepezil 10 mg: Par. in this arm received donepezil 5 mg capsule along with dummy RSGXR tablet once daily for the first 4W of treatment. From Visit 4 (W4) onwards, these par. received donepezil 10 mg capsule along with dummy RSGXR tablet once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
Period: Overall Study
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Started | 165 | 166 | 165 | 83
Completed | 131 | 135 | 127 | 55
Not Completed | 34 | 31 | 38 | 28
Not completed — Adverse Event | 10 | 8 | 10 | 11
Not completed — Lost to Follow-up | 3 | 6 | 1 | 4
Not completed — Protocol Violation | 3 | 1 | 3 | 3
Not completed — Withdrawal by Subject | 10 | 12 | 15 | 5
Not completed — Sponsor terminated study | 0 | 1 | 0 | 0
Not completed — Non-compliance | 4 | 0 | 1 | 3
Not completed — Par. did not returned to visit | 1 | 0 | 0 | 1
Not completed — Follow-Up visit not possible | 1 | 0 | 0 | 0
Not completed — Prohibited medication used for SAE | 1 | 0 | 0 | 0
Not completed — Death of par. | 1 | 0 | 1 | 0
Not completed — Visit 7 exceed the visit window | 0 | 1 | 0 | 0
Not completed — Medical monitor terminated par. | 0 | 1 | 0 | 0
Not completed — Mental status of par. was | 0 | 1 | 0 | 0
Not completed — Worsening of AD | 0 | 0 | 1 | 0
Not completed — Excluded for concerning QTc value | 0 | 0 | 1 | 0
Not completed — Insufficient AD documentation | 0 | 0 | 1 | 0
Not completed — High MMSE scores | 0 | 0 | 1 | 0
Not completed — Deterioration of cognitive status | 0 | 0 | 1 | 0
Not completed — Serious adverse event | 0 | 0 | 1 | 0
Not completed — Excluded for heart insufficiency | 0 | 0 | 1 | 0
Not completed — Raised Creatinine Value | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was used and consist of all par. randomized to treatment, who have taken at least one dose of study medication and who have at least one post baseline efficacy assessment. The ITT population included 553 participants.
Groups:
- RSG XR 2 mg: Par. in this arm received RSGXR 2 milligram (mg) tablet along with dummy donepezil capsule once daily for 24W. For par. in this arm, the dosage were remain constant throughout the 24W treatment period. Study treatment were taken in the evening with or without food.
- Total: Total of all reporting groups
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg | Total
Number analyzed (Participants) | 159 | 162 | 156 | 76 | 553
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data are presented for intention-to-Treat (ITT) population which defined as par. randomized to treatment, who have taken at least one dose of study medication and who have at least one post baseline efficacy assessment (Alzheimer's Disease Assessment Scale - Cognitive subscale [ADAS-Cog] or Clinician's Interview-Based Impression of Change Plus [CIBIC+]).
  Years | 72.5 (8.56) | 71.7 (7.91) | 72.6 (8.63) | 72.9 (7.97) | 72.4 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants] — ITT Population
  Participants
    Female | 95 | 103 | 101 | 48 | 347
    Male | 64 | 59 | 55 | 28 | 206
Race (NIH/OMB) [Count of Participants; unit: Participants] — ITT Population
  Participants
    American Indian or Alaska Native | 1 | 1 | 2 | 0 | 4
    Asian | 33 | 50 | 37 | 14 | 134
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 1 | 2 | 3 | 7
    White | 123 | 109 | 112 | 57 | 401
    More than one race | 1 | 1 | 3 | 2 | 7
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (W0) in Mean ADAS-Cog Total Score at W24 as a Function of APOE e4 Status in Apolipoprotein epsilon4 (APOE e4) Negative Cohort
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Items were evaluated by tests and clinician ratings on a 5-point scale. Scores ranged from 0-70 with higher scores indicates more dysfunction. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline is defined as value at W0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. A hierarchical testing procedure was used to control for the two rosiglitazone dose groups and the three genetic subgroups. There was no adjustment for the donepezil versus placebo comparisons, which were included to assess the sensitivity of the trial to detect a treatment effect.
Time Frame: Baseline (W0) and W24
Population: ITT Population. Only those par. available at the indicated time points were analyzed. These comparisons were conducted for APOE e4 negative (neg) par. (e2/e2, e2/e3, and e3/e3) cohort
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Placebo: Par. randomized to this arm received RSG placebo tablet along with dummy donepezil capsule once daily for 24W. For par. in this arm, the dosage were remain constant throughout the 24W treatment period. Study treatment were taken in the evening with or without food.
- RSG XR 2 mg: Par. randomized to this arm received RSGXR 2 milligram (mg) tablet along with dummy donepezil capsule once daily for 24W. For par. in this arm, the dosage were remain constant throughout the 24W treatment period. Study treatment were taken in the evening with or without food.
- RSG XR 8 mg: Par. randomized to this arm received RSGXR 4 mg tablet along with dummy donepezil capsule once daily for the first 4 weeks of treatment. From Visit 4 (Week 4) onwards, these par. received 8 mg RSGXR tablet along with dummy donepezil capsule once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
- Donepezil 10 mg: Par. randomized to this arm received donepezil 5 mg capsule along with dummy RSGXR tablet once daily for the first 4 weeks of treatment. From Visit 4 (Week 4) onwards, these par. received donepezil 10 mg capsule along with dummy RSGXR tablet once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 63 | 69 | 65 | 28
Score on a scale | 1.6 (0.78) | -0.2 (0.67) | 0.6 (0.67) | 0.9 (1.16)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.074, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg in APOE e4 neg cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.8 to 0.2] — Difference in adjusted least square means was shown (Active treatment minus Placebo); n = Number of par. with evaluable data
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.338, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg in APOE e4 neg cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-3.0 to 1.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.602, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10mg in APOE e4 neg cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.5 to 2.1] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline (W0) in Mean ADAS-Cog Total Score at W24 as a Function of APOE e4 Status in All Except e4/e4's Cohort
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Items were evaluated by tests and clinician ratings on a 5-point scale. Scores ranged from 0-70 with higher scores indicates more dysfunction. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline is defined as value at W0. Estimated value was calculated by Active treatment minus Placebo. A hierarchical testing procedure was used to control for the two rosiglitazone dose groups and the three genetic subgroups. There was no adjustment for the donepezil versus placebo comparisons, which were included to assess the sensitivity of the trial to detect a treatment effect.
Time Frame: Baseline (W0) and W24
Population: ITT Population. Only those par. available at the indicated time points were analyzed. These comparisons were conducted in all except e4/e4's: comprised of APOE e4 neg par. (e2/e2, e2/e3, and e3/e3) and APOE e4 heterozygote par. (e2/e4, e3/e4)
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 117 | 115 | 112 | 49
Score on a scale | 1.5 (0.58) | 0.3 (0.54) | 0.7 (0.57) | -0.1 (0.79)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.131, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg in All except e4/e4's cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.7 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.315, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg in All except e4/e4's cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.4 to 0.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.105, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg in All except e4/e4's cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.5 to 0.3] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline (W0) in Mean ADAS-Cog Total Score at W24 as a Function of APOE e4 Status in Full Population Cohort
Description: as for outcome 2
Time Frame: Baseline (W0) and W24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 131 | 130 | 125 | 56
Score on a scale | 2.0 (0.56) | 1.2 (0.53) | 1.2 (0.55) | 0.6 (0.74)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.272, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.2 to 0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.297, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.2 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.131, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.1 to 0.4]

4. Primary Outcome: Change From Baseline (W0) in Mean CIBIC+ Global Functioning Total Score at W24 as a Function of APOE e4 Status in APOE4 Negative Cohort
Description: The CIBIC+ assessment comprised of a 7-point rating of severity (at baseline) and change (at indicated time points). It was rated on a scale of 1 to 7 as 1: markedly improved, 2.: moderately improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: moderately worse and 7: markedly worse; higher score means greater dysfunction. It was based on interviews with the par. and caregiver by an independent rater. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived. Estimated value was calculated by Active treatment minus Placebo. A hierarchical testing procedure was used to control for the two rosiglitazone dose groups and the three genetic subgroups. There was no adjustment for the donepezil versus placebo comparisons, which were included to assess the sensitivity of the trial to detect a treatment effect.
Time Frame: Baseline (W0) and W24
Population: ITT Population. Only those par. available at the indicated time points were analyzed. These comparisons were conducted in APOE e4 negative (neg) par. (e2/e2, e2/e3, and e3/e3).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 63 | 71 | 66 | 28
Score on a scale | 4.2 (0.14) | 4.2 (0.12) | 4.1 (0.11) | 3.9 (0.22)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.663, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg in APOE e4 neg cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.891, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg in APOE e4 neg cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.414, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg in APOE e4 neg cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.7 to 0.3] — Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix

5. Primary Outcome: Change From Baseline (W0) in Mean CIBIC+ Global Functioning Total Score at W24 as a Function of APOE e4 Status in All Except e4/e4's Cohort
Description: as for outcome 4
Time Frame: Baseline (W0) and W24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 117 | 117 | 114 | 49
Score on a scale | 4.3 (0.10) | 4.3 (0.10) | 4.1 (0.10) | 3.8 (0.17)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.913, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg in All except e4/e4's cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.276, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg in All except e4/e4's cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.025, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg in All except e4/e4's cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.1] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Change From Baseline (W0) in Mean CIBIC+ Global Functioning Total Score at W24 as a Function of APOE e4 Status in Full Population Cohort
Description: as for outcome 4
Time Frame: Baseline (W0) and W24
Population: ITT Population. Only those par. available at the indicated time points were analyzed. These comparisons were conducted in full population.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 131 | 133 | 127 | 56
Score on a scale | 4.3 (0.09) | 4.3 (0.09) | 4.2 (0.10) | 3.8 (0.16)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.939, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.307, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.009, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.1] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline (W0) in Mean ADAS-Cog Total Score at W8, W16, W24
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a 5-point scale. Scores ranged from 0-70 with higher scores indicating greater dysfunction. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline is defined as value at W0. Endpoint treatment differences were adjusted to take account of missing data. It was evaluated at Baseline, W8, W16 and W24.
Time Frame: Baseline (W0) and up to W24
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented as n=x,x,x,x in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  ADAS-Cog, W8, n=153, 155,147,67 | 0.4 (0.42) | -0.5 (0.45) | 0.5 (0.43) | -0.3 (0.63)
  ADAS-Cog, W16, n=143,145,132,62 | 0.5 (0.46) | 0.6 (0.49) | 1.3 (0.45) | -1.1 (0.80)
  ADAS-Cog, W24, n=131, 130,125,156 | 2.0 (0.56) | 1.2 (0.53) | 1.2 (0.55) | 0.6 (0.74)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.116, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.0 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.816, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.9 to 1.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.318, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.1 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.839, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg in at Week 16 Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.1 to 1.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.165, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.3 to 2.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.073, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.4 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.272, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.2 to 0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.297, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.2 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.131, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.1 to 0.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline (W0) in Mean CIBIC+ Global Functioning Total Score at W8, W16, W24
Description: The CIBIC+ assessment comprised of a 7-point rating of severity (at baseline) and change (at indicated time points). It was rated on a scale of 1 to 7 as 1: markedly improved, 2.: moderately improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: moderately worse and 7: markedly worse; higher score means more dysfunction. The scale was based on interviews with the par. and caregiver and was completed by an independent rater. It required separate structured 15-20 minute interviews with the par. and caregiver. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived. It was evaluated at Baseline, W8, W16 and W24.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  CIBIC+, W8, n=150, 156,147,67 | 4.1 (0.07) | 3.9 (0.08) | 4.1 (0.08) | 3.9 (0.12)
  CIBIC+, W16, n=144,145,127,61 | 4.2 (0.08) | 4.0 (0.08) | 4.1 (0.09) | 3.8 (0.14)
  CIBIC+, W24, n=131,133, 127, 56 | 4.3 (0.09) | 4.3 (0.09) | 4.2 (0.10) | 3.8 (0.16)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.133, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.958, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.085, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.102, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.380, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.006, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.939, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.307, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.009, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.1] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline (W0) in Mean Neuropsychiatric Inventory (NPI) Total Score at W8, W16, W24
Description: The NPI assessed behavioral disturbances comprises 10 dimensions: delusions, hallucinations, dysphoria, apathy, euphoria, disinhibition, aggressiveness and agitation, irritability, anxiety and aberrant motor activity. The par. caregiver asked about behavior in the par. If "Yes", the informant then rates both the severity on a 3-point scale, 1: mild to 3: severe (total range: 0-36) and the frequency using a 4-point scale, 1: occasionally to 4: very frequently. The total domain score was frequency × severity. The distress was scored on 5-point scale, 0: no distress to 5 - very severe or extreme. A total NPI score can be calculated by adding all domain scores together; NPI total score: from 0-144 and NPI distress score: from 0-60, all with higher scores indicating more severe behavioral disturbance. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0.
Time Frame: Baseline (W0) and up to W24
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented as n=x,x,x,x in the category titles). Endpoint treatment differences which were adjusted to take account of missing data are derived.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- RSG XR 8 mg: Par. in this arm received RSGXR 4 mg tablet along with dummy donepezil capsule once daily for the first 4 weeks of treatment. From Visit 4 (Week 4) onwards, these par. received 8 mg RSGXR tablet along with dummy donepezil capsule once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
- Donepezil 10 mg: Par. in this arm received donepezil 5 mg capsule along with dummy RSGXR tablet once daily for the first 4 weeks of treatment. From Visit 4 (Week 4) onwards, these par. received donepezil 10 mg capsule along with dummy RSGXR tablet once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  NPI, W8, n=146,151,144,65 | 0.2 (0.59) | 0.1 (0.63) | 0.5 (0.81) | -0.1 (0.87)
  NPI, W16, n=139,142,131,59 | -0.1 (0.69) | -0.0 (0.69) | -0.1 (0.90) | 0.5 (0.97)
  NPI, W24, n=129,133,127,55 | 1.2 (1.04) | 1.6 (0.74) | 1.1 (1.01) | -0.6 (1.12)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.957, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.6 to 1.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.693, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.4 to 2.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.798, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.2 to 1.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.958, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.7 to 1.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.998, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-2.1 to 2.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.639, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.5, 95% CI [-1.7 to 2.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.797, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.1 to 2.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.942, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.9 to 2.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.213, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.8 to 1.1] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline (W0) in Mean Disability Assessment for Dementia (DAD) Scale Total Score at W8, W16, W24
Description: The DAD, assessed the ability of a par. to execute basic and instrumental activities of daily living (ADL) and leisure activities. The scale consists of 40 questions assessing basic and instrumental ADLs. This scale assesses a participants' ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item was scored as yes: 1, no: 0 and N/A: not applicable. Higher scores indicate less disability with a score of 100 indicating no disability and 0 indicating no functional ability. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. The percentage score was calculated as (DAD total score/total number of applicable items) multiplied by 100. Endpoint treatment differences which were adjusted to take account of missing data are derived.
Time Frame: Baseline (W0) and up to W24
Population: ITT Population. Only those par. available at the specified time points were analyzed (represented as n=x,x,x,x in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  DAD, W8, n=147,152, 144, 65 | -0.8 (0.80) | -0.6 (0.94) | -0.3 (0.78) | 0.5 (1.00)
  DAD, W16, n=141,143,131,59 | -2.6 (0.98) | -1.7 (1.07) | -1.7 (1.05) | 1.1 (1.40)
  DAD, W24, n=129,133,127,55 | -3.7 (0.97) | -2.4 (1.21) | -3.8 (1.19) | -0.2 (1.81)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.919, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.1 to 2.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.649, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.5 to 2.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.279, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-1.1 to 3.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.498, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-1.8 to 3.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.489, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg in at Week 16 Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-1.7 to 3.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.024, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [0.5 to 7.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.385, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-1.6 to 4.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.944, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-3.0 to 2.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.078, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-0.4 to 7.5] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change From Baseline (W0) in Mean Short Term Memory Assessment Total Score (ADAS-Cog Q1 Plus Q7) at W8, W16, W24
Description: Change from Baseline in short term memory assessment score was assessed from a combined analysis of items 1 (word recall task) and 7 (word recognition task) of ADAS-Cog scale. Word recall task consist of the participants score was the mean number of words not recalled on three trials (maximum score 10) and word recognition task, to score this item the number of incorrect responses was counted (maximum error score was 12). Higher score indicating greater dysfunction. Total score is sum of individual score. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  ADAS-Cog Q1 plus Q7, W8, n=152,155,146,67 | 0.1 (0.25) | -0.1 (0.27) | 0.5 (0.25) | -0.4 (0.40)
  ADAS-Cog Q1 plus Q7, W16, n=143,143,130,62 | 0.1 (0.27) | 0.6 (0.26) | 0.8 (0.24) | -0.6 (0.45)
  ADAS-Cog Q1 plus Q7, W24, n=131,128,123,56 | 0.7 (0.27) | 0.3 (0.30) | 0.6 (0.29) | 0.2 (0.43)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.635, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.8 to 0.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.194, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.2 to 1.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.325, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 8 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.3 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.109, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.1 to 1.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.032, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [0.1 to 1.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.189, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 16 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.7 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.288, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.819, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.306, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.5 to 0.5] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline (W0) in Mean European Quality of Life -5 Dimensions Proxy Version (EQ-5D Proxy) Total Score at W12, W24 Assessed by Utility
Description: The EQ-5D Proxy was a 2 part scale used to assess the quality of life and utility benefit. The data for Part 1 is presented. It is a 5 dimensional Health State Classification. Caregivers were asked to respond as they feel the par. would on dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Answers to each question were recorded on a 3-point scale which indicates the level of impairment (level 1= no problem; level 2=some or moderate problem(s) and level 3=unable, or extreme problem with higher scores indicating greater dysfunction. EQ-5D Proxy assessments was performed at Baseline, W12 and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  EQ-5D Proxy Utility, W12, n=141,146, 135, 62 | -0.02 (0.017) | 0.00 (0.016) | 0.01 (0.016) | 0.01 (0.021)
  EQ-5D Proxy Utility, W24, n=128, 130, 125, 55 | -0.02 (0.017) | 0.02 (0.016) | -0.02 (0.019) | 0.00 (0.018)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.199, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.094, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.01 to 0.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.187, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.02 to 0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.134, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.958, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.05 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.374, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.07] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline (W0) in Mean European Quality of Life -5 Dimensions Proxy Version (EQ-5D Proxy) Total Score at W12, W24 Assessed by Thermometer (Visual Analog Scale [VAS])
Description: The EQ-5D Proxy is a 2 part scale used to assess the quality of life and utility benefit. The data for Part 2 is presented. It is a the visual analogue scale Thermometer which assessed caregiver's impression of par. overall health. The Thermometer has endpoints of 100 (best imaginable health state) and 0 (worst imaginable health state). EQ-5D Proxy assessments was performed at Baseline, W12 and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  EQ-5D Proxy Thermometer, W12, n=141, 146, 135, 62 | 1.4 (1.35) | 0.3 (1.37) | 1.7 (1.41) | -2.6 (2.41)
  EQ-5D Proxy Thermometer, W24, n=128, 130, 126, 55 | 1.9 (1.56) | -0.7 (1.52) | 0.2 (1.71) | 1.5 (2.40)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.493, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-4.6 to 2.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.883, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-3.2 to 3.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.130, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-9.3 to 1.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.198, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-6.6 to 1.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.441, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-5.9 to 2.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.898, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-5.8 to 5.1] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Time Spent Caring for Basic and Instrumental Activities Resource Utilization in Dementia (RUD) Scale at W12 and W24
Description: The RUD instrument was developed as a comprehensive tool to assess the amount of resource use among demented par. RUD assess both formal and informal resource use of the par. and the primary caregiver, making it possible to calculate costs from a societal perspective. Q1 relates to assisting par. with basic activities of daily living and Q2 relates to instrumental activities of daily living. The assessments was performed at Baseline, W12 and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Hours
  RUD Q1, W12, n=141, 149, 137, 69 | 2.3 (43.31) | 4.5 (81.21) | -9.8 (77.44) | -5.7 (70.19)
  RUD Q1, W24, n=128, 133, 127, 55 | 19.4 (109.41) | -0.6 (58.72) | -2.7 (86.26) | 3.7 (19.26)
  RUD Q2, W12, n=141, 149, 137, 62 | 13.7 (73.94) | 9.0 (60.54) | 4.9 (80.97) | -5.3 (56.50)
  RUD Q2, W24, n=128, 133, 127, 55 | 17.1 (75.45) | 9.7 (47.96) | 11.6 (107.52) | 1.1 (61.49)

15. Secondary Outcome: Change From Baseline (W0) in Alzheimer's Carer's Quality of Life Instrument (ACQLI) Score at W12 and W24.
Description: The ACQLI was an assessment of caregiver quality of life. This instrument consists of 30 questions exploring various aspects of carer's quality of life. Each of the questions had a two point response and the 30 questions were summed to provide a total score. Items are assumed to be unidimensional (i.e., represent a single variable) and are scored 0/1 (false/true) before summation into a total score with a 0-30 range. To ease comparisons between scales, ACQLI scores were transformed to range between 0-100 (100: worse). The assessments was performed at Baseline, W12 and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 159 | 162 | 156 | 76
Score on a scale
  ACQLI, W12, n=141, 148, 137, 60 | 0.5 (0.38) | -0.6 (0.41) | -0.1 (0.46) | 0.5 (0.50)
  ACQLI, W24, n=128, 132, 126, 54 | 0.6 (0.45) | -0.2 (0.49) | 0.0 (0.54) | -0.0 (0.69)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.027, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.1 to -0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.278, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.6 to 0.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.993, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 12 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.2 to 1.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.196, Mixed model for repeated measures — Comparison between Placebo and RSG XR 2 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.0 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.353, Mixed model for repeated measures — Comparison between Placebo and RSG XR 8 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.9 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.427, Mixed model for repeated measures — Comparison between Placebo and Donepezil 10 mg at Week 24 in Full population cohort; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-2.2 to 0.9] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Change From Baseline (W0) in Mini Mental State Examination (MMSE) Total Score at W24.
Description: The MMSE consists of 11 tests of orientation, memory (recent and immediate), concentration, language and praxis. Scores range from 0 to 30, with lower scores indicating greater cognitive impairment. The scale is completed by the investigator, based on the performance of the par. and takes approximately 5 to 10 minutes to administer. The assessments was performed at Baseline and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived
Time Frame: Baseline (W0) and W24
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 131 | 133 | 127 | 56
Score on a scale | -0.5 (0.27) | -0.6 (0.27) | -0.7 (0.28) | 0.4 (0.38)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.886, ANCOVA; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.7 to 0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.710, ANCOVA; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.030, ANCOVA; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [0.1 to 1.8] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Change From Baseline (W0) in Glycosylated Hemoglobin (HbA1c) at W24.
Description: The blood sample was collected for assessments of HbA1c levels at Baseline and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0. Endpoint treatment differences which were adjusted to take account of missing data are derived.
Time Frame: Baseline (W0) and W24
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Groups:
- Donepezil 10 mg: Par. in this arm received donepezil 5 mg capsule along with dummy RSGXR tablet once daily for the first 4Wof treatment. From Visit 4 (W4) onwards, these par. received donepezil 10 mg capsule along with dummy RSGXR tablet once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 123 | 120 | 117 | 52
Percentage (%) | 0.1 (0.05) | 0.2 (0.05) | 0.1 (0.05) | 0.1 (0.07)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2 mg; Test type: Superiority or Other; p = 0.139, ANCOVA; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.0 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8 mg; Test type: Superiority or Other; p = 0.846, ANCOVA; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Donepezil 10 mg; Test type: Superiority or Other; p = 0.864, ANCOVA; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.1 to 0.2] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Number of Participants With Adverse Events Defined by Severity
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE included significant or unexpected worsening or exacerbation of the condition/indication under study, exacerbation of a chronic or intermittent pre-existing condition, new conditions detected or diagnosed, signs, symptoms, or the clinical sequelae of a suspected overdose of either investigational product or a concurrent medication. Number of participants with any AE and as per severity were reported. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: Up to W24
Population: Safety population: This included all par. randomized to treatment who have taken at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
Participants
  Any AE | 62 | 60 | 69 | 42
  Mild AE | 32 | 35 | 37 | 22
  Moderate AE | 25 | 22 | 30 | 15
  Severe AE | 5 | 3 | 2 | 5

19. Secondary Outcome: Number of Participants With Systolic and Diastolic Blood Pressure (SBP and DBP), Heart Rate (HR) and Weight Values of Potential Clinical Concern (PCC) Any Time on Treatment (ATOT).
Description: SBP, DBP and HR of par. were recorded in sitting posture as vital signs, while body weight was measured without shoes and wearing light clothing at each visit. The blood pressure (BP) and HR values were identified as of PCC if the vales were out of the reference range (for SBP, 90 to 140 millimeters of mercury (mmHg), DBP, 50 to 90 mmHg, and HR >100 or <50 beats per minute [bpm]) or meet a change from Baseline criterion. For SBP it was increase from Baseline (high) if increased by more than or equal to (>=) 40 mmHg; decrease from Baseline (low) if decreased by >=30 mmHg. For DBP, increase from Baseline (high) if increased by >=30 mmHg; decrease from Baseline (low) if decreased by >=20 mmHg. For HR, increase from Baseline (high) if increased by >=30 bpm; decrease from Baseline (low) if decreased by >=30 bpm. For weight, increase from Baseline (high) if increased by >=7%; decrease from Baseline (low) if decreased by >=7%. Baseline was defined as value at W0.
Time Frame: Up to W24
Population: Safety Population. Only those par. available at the specified time points were analyzed (represented as n=x,x,x,x in the category titles).
Measure: Number; unit: Participants
Groups:
- Donepezil 10 mg: Par.in this arm received donepezil 5 mg capsule along with dummy RSGXR tablet once daily for the first 4W of treatment. From Visit 4 (W4) onwards, these par. received donepezil 10 mg capsule along with dummy RSGXR tablet once daily for the remaining 20W of double-blind treatment. Study treatment were taken in the evening with or without food.
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 160 | 162 | 154 | 79
Participants
  SBP, >140 or <90 | 52 | 61 | 41 | 24
  SBP, Increase from Baseline >=40 | 1 | 3 | 3 | 3
  SBP, Decrease from Baseline >=30 | 7 | 9 | 15 | 6
  DBP, >90 or <50 | 17 | 16 | 13 | 8
  DBP, Increase from Baseline >=30 | 4 | 1 | 1 | 1
  DBP, Decrease from Baseline >=20 | 8 | 12 | 25 | 8
  HR, >100 or <50 | 2 | 4 | 4 | 2
  HR, Increase from Baseline >=30 | 1 | 3 | 3 | 1
  HR, Decrease from Baseline >=30 | 3 | 0 | 0 | 1
  Weight, Increase from Baseline >=7% | 9 | 21 | 25 | 1
  Weight, Decrease from Baseline >=7% | 7 | 4 | 3 | 5

20. Secondary Outcome: Change From Baseline (W0) in 12-lead Electrocardiogram (ECG)
Description: Triplicate 12-lead ECG measures was obtained digitally, approximately one minute apart after the par. had rested in the supine position in a quiet room (no TV, minimal talking) for at least 10 minutes. Conduction intervals from the 12-lead ECGs were manually read and confirmed by an external cardiologist/vendor. The ECG parameters includes PR interval, QRS duration, QT - uncorrected interval, QTc Bazett (QTcB), QTc Fridericia (QTcF) and RR interval of Central Cardiologist are reported. The assessments was performed at Baseline and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Screening/Visit 1/W-6.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: milliseconds (MSEC)
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
milliseconds (MSEC)
  PR Interval, n=16,11, 14, 4 | 2.2 (14.39) | 6.9 (30.44) | 6.0 (19.98) | -5.5 (8.50)
  QRS Duration, n=17, 11, 14, 5 | 1.1 (8.28) | 0.7 (5.50) | 3.6 (6.14) | 0.9 (9.04)
  QT Interval, n=17, 11, 14, 5 | 5.3 (27.69) | 15.6 (25.06) | 19.8 (22.17) | 15.9 (22.57)
  QTcB, n=17, 11, 14, 5 | 10.2 (18.21) | 7.1 (22.69) | 20.0 (13.54) | -0.2 (17.22)
  QTcF, n=17, 11, 14, 5 | 8.1 (17.12) | 10.0 (21.47) | 20.1 (12.71) | 4.9 (15.50)
  RR Interval | -12.3 (107.35) | 43.8 (89.52) | -0.5 (107.49) | 76.5 (109.43)

21. Secondary Outcome: Change From Baseline (W0) in Heart Rate (HR) Measured From 12-lead Electrocardiogram (ECG)
Description: Triplicate 12-lead ECG measures was obtained digitally, approximately one minute apart after the par. had rested in the supine position in a quiet room (no TV, minimal talking) for at least 10 minutes. Conduction intervals from the 12-lead ECGs were manually read and confirmed by an external cardiologist/vendor. The ECG HR of Central Cardiologist reported. The assessments was performed at Baseline and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Screening/Visit 1/W-6.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 17 | 11 | 14 | 5
Beats per minute | 2.1 (12.08) | -2.8 (7.77) | -0.3 (8.39) | -4.7 (9.23)

22. Secondary Outcome: Change From Baseline (W0) in Body Weight
Description: Body weight will be measured at all visits, without shoes and wearing light clothing. The assessments was performed at Baseline, W4, W8, W12, W16, and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
Kilogram (Kg)
  Week 4, n=160, 161, 153, 79 | 0.1 (1.59) | 0.4 (1.76) | 0.3 (1.61) | -0.1 (1.39)
  Week 8, n=150, 157, 147, 66 | -0.0 (2.56) | 0.5 (1.73) | 0.8 (2.16) | -0.4 (1.46)
  Week 12, n=143, 149, 136, 61 | 0.0 (2.12) | 0.6 (2.06) | 0.9 (2.03) | -0.9 (1.71)
  Week 16, n=143, 146, 132, 61 | -0.0 (2.05) | 0.7 (2.20) | 1.1 (2.08) | -1.0 (2.05)
  Week 24, 133, 132, 125, 55 | -0.3 (2.53) | 0.8 (2.63) | 0.8 (2.54) | -0.8 (2.28)

23. Secondary Outcome: Change From Baseline (W0) in Hemoglobin
Description: Hematology parameters were assessed at Baseline, W4, W12 and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
Grams per liter (G/L)
  Week 4, n=152, 152, 138, 76 | 0.1 (5.84) | -2.8 (7.04) | -3.9 (7.57) | -0.4 (6.03)
  Week 12, n=132, 142, 132, 60 | -0.2 (6.55) | -4.5 (8.65) | -10.5 (8.67) | -0.6 (6.59)
  Week 24, n=128, 124, 115, 54 | -1.3 (7.54) | -4.2 (8.34) | -11.9 (10.58) | 0.2 (6.51)

24. Secondary Outcome: Change From Baseline (W0) in Hematocrit
Description: as for outcome 23
Time Frame: Baseline (W0) and Up to W24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
Percentage of red blood cells in blood
  Week 4, n=152, 152, 138, 76 | -0.0011 (0.01886) | -0.0088 (0.02285) | -0.0125 (0.02322) | -0.0024 (0.01829)
  Week 12, n=132, 142, 132, 60 | -0.0007 (0.02137) | -0.0152 (0.02813) | -0.0316 (0.02629) | -0.0055 (0.01932)
  Week 24, n=128, 124, 115, 54 | -0.0010 (0.02500) | -0.0123 (0.02304) | -0.0326 (0.03195) | -0.0001 (0.02135)

25. Secondary Outcome: Change From Baseline (W0) in Periodic HbA1c Assessment
Description: HbA1c assessment was performed par. with type 2 diabetes mellitus or HbA1c >=6.5% at Screening only. HbA1c levels were assessed at Baseline, W12 and W24. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at W0.
Time Frame: Baseline (W0) and up to W24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
Percentage
  Week 12, n=48, 46, 38, 22 | -0.1 (0.56) | 0.2 (0.62) | 0.1 (0.41) | -0.2 (0.81)
  Week 24, n=123, 120, 117, 52 | 0.1 (0.52) | 0.2 (0.66) | 0.1 (0.52) | 0.0 (0.56)

26. Secondary Outcome: Number of Par. With Hematology Data of Potential Clinical Concern Any Time on Treatment
Description: Haematology parameters were identified as of PCC (high [H], low [L]), if the values were out of the reference range (RR). The range for parameters was: platelet (100AV-500AV), red blood cell (RBC, 0.8-1.2), hemoglobin (L: female [F]:10, male [M]:11; H: F:16.5-AV, M:18), hematocrit (0.8-1.2), white blood cell (WBC, 3-15), neutrophils (0.75-1.5), lymphocytes (0.75-1.5), monocytes (0.75-2), eosinophils (none-2), basophils (none-2), mean corpuscle volume (MCV, 0.8-1.2), mean corpuscular hemoglobin (MCH, 0.8-1.2), mean corpuscular hemoglobin concentration (MCHC, 0.8-1.2), red cell distribution width (RDW, 0.8-1.2). Data for mean platelet volume (reference range not established) not reported
Time Frame: Up to W24
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
Participants
  Eosinophils H, n=156, 161, 151, 72 | 2 | 0 | 1 | 0
  Hematocrit H, n=157, 161,151, 76 | 0 | 1 | 0 | 0
  Hematocrit L, n=157, 161,151, 76 | 0 | 0 | 1 | 0
  Hemoglobin H, n=157, 161,151, 76 | 0 | 2 | 0 | 0
  Hemoglobin L, n=157, 161,151, 76 | 0 | 3 | 8 | 0
  Lymphocytes L, n=156, 161,151, 76 | 2 | 2 | 2 | 0
  MCH H, n=157, 161,151, 76 | 0 | 0 | 0 | 1
  MCH L, n=157, 161,151, 76 | 0 | 1 | 0 | 0
  MCV L, n=156, 161,151, 76 | 0 | 0 | 0 | 1
  Monocytes H, n=156, 161,151, 76 | 0 | 0 | 0 | 1
  Monocytes L, n=156, 161,151, 76 | 9 | 10 | 15 | 4
  Platelet H, n=157, 160,150, 76 | 1 | 0 | 0 | 0
  Platelet L, n=157, 160,150, 76 | 2 | 1 | 0 | 0
  RDW H, n=157, 161,151, 76 | 4 | 6 | 10 | 1
  RBC L, n=157, 161,151, 76 | 0 | 1 | 1 | 1
  Total neutrophil H, n=156, 161, 151, 76 | 0 | 0 | 1 | 1
  Total neutrophil L, n=156, 161, 151, 76 | 2 | 5 | 7 | 3
  WBC H, n=157, 161,151, 76 | 0 | 0 | 1 | 1
  WBC L, n=157, 161,151, 76 | 4 | 4 | 7 | 0

27. Secondary Outcome: Number of Par. With Clinical Chemistry Values of Potential Clinical Concern Any Time on Treatment
Description: Clinical chemistry parameters were identified as of PCC (H, L), if values were out of RR: Alanine aminotransferase (ALT, none-120 [250% upper limit of RR, ULRR]), Albumin (0.75-2), Aspartate aminotransferase (AST,none-105 (3-64y), 137.5 (65+y), >250%ULRR), Alkaline phosphatase (ALP,none-312.5 (20+y), >250%ULRR), blood urea nitrogen (BUN)/Creatinine ratio (none-1.25), BUN (none-11), Chloride (80-115), Calcium (0.75-1.25), Carbon dioxide (CO2, 15-40) content, Creatinine (22, <50% lower limit of RR [LLRR]-155, >125%ULRR), Creatine phosphokinase (CPK, none-1.25), Gamma glutamyl transferase (GGT,none-2.5), Glucose (3.6-7.8), High density lipoprotein (HDL,0.65-none), Lactate dehydrogenase (LDH,none-1.25), Low density lipoprotein (LDL,none-2), Magnesium (0.5-2), Potassium (3-5.5), Phosphorus inorganic (0.5-1.5), Sodium (130-150), Total protein (0.8-1.5), Total cholesterol (none-1.25), Total bilirubin (none-1.95), Triglycerides (none-9). Data for Creatinine clearance not reported.
Time Frame: Up to W24
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
Number analyzed (Participants) | 165 | 166 | 165 | 83
Participants
  ALT H, n=156, 162, 151, 77 | 2 | 0 | 0 | 0
  AST H, n=156, 162, 151, 77 | 2 | 0 | 0 | 0
  BUN/Creatinine ratio H, n=156, 162, 151, 77 | 8 | 8 | 19 | 9
  Cholesterol H, n=141, 148, 137, 62 | 7 | 17 | 29 | 1
  Creatinine H, n=156, 162, 151, 77 | 5 | 1 | 4 | 3
  CPK H, n=156, 162, 151, 77 | 5 | 13 | 11 | 5
  GGT H, n=156, 162, 151, 77 | 2 | 1 | 0 | 1
  Glucose H, n=156, 162, 151, 77 | 12 | 19 | 9 | 8
  Glucose L, n=156, 162, 151, 77 | 3 | 5 | 4 | 1
  LDL H, n=141, 147, 136, 62 | 36 | 51 | 55 | 10
  Phosphorus L, n=156, 162, 151, 77 | 0 | 0 | 1 | 0
  Potassium H, n=156, 162, 150, 77 | 4 | 2 | 2 | 2
  Sodium H, n=156, 162, 151, 77 | 0 | 0 | 0 | 1
  Sodium L, n=156, 162, 151, 77 | 0 | 0 | 1 | 2
  BUN H, n=156, 162, 151, 77 | 7 | 5 | 12 | 5
  Total Bilirubin H, n=156, 162, 151, 77 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication up to W24.
Description: The safety population (full population cohort) was used.
Arm/Group | Placebo | RSG XR 2 mg | RSG XR 8 mg | Donepezil 10 mg
All-Cause Mortality (participants affected / at risk) | 1/165 | 0/166 | 1/165 | 0/83
Serious Adverse Events (participants affected / at risk) | 10/165 | 7/166 | 8/165 | 6/83
Other Adverse Events (participants affected / at risk) | 13/165 | 25/166 | 30/165 | 11/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | RSG XR 2 mg (N=166) | RSG XR 8 mg (N=165) | Donepezil 10 mg (N=83)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Discomfort (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | RSG XR 2 mg (N=166) | RSG XR 8 mg (N=165) | Donepezil 10 mg (N=83)
Oedema peripheral (General disorders) | 9 | 6 | 24 | 3
Nasopharyngitis (Infections and infestations) | 4 | 11 | 4 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 9 | 1 | 2
Headache (Nervous system disorders) | 0 | 2 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.